CLINICAL TRIAL: NCT06891417
Title: A Phase 1/2, Randomized, Placebo-controlled, Multi-arm, Dose-finding Study to Evaluate the Safety, Immunogenicity, and Efficacy of a Chlamydia Trachomatis mRNA Vaccine Candidate in Adults Aged 18 to 29 Years
Brief Title: Phase 1/2 Study of Chlamydia Trachomatis mRNA Vaccine in Adults Aged 18 to 29 Years
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: VAV00023; U1111-1308-7349 (Other: WHO ICTRP)
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Chlamydia Trachomatis Immunization
Keywords: Chlamydia
MeSH Terms: conditions — Chlamydia Infections

STUDY DESIGN:
Intervention Model Description: Sequential (Phase 1) / parallel (Phase 2), dose finding, multi center
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sentinel Cohorts: modified double-blind
  * Investigator, participants, and laboratory personnel will be blinded
  * Clinical site staff preparing / administering the study vaccines will be unblinded
  * Sponsor study staff involved in the early safety data review (ESDR) will be unblinded at the time of the ESDR Main Cohort: modified double-blind
  * Investigator, participants, laboratory personnel, and Sponsor study staff will be blinded
  * Only clinical site staff preparing / administering the study vaccines will be unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- Sentinel Cohort A Group 1: Chlamydia trachomatis Seronegative (Experimental): Participants will receive three low dose injections of Chlamydia mRNA Vaccine
  Interventions: Biological: Chlamydia mRNA Vaccine
- Sentinel Cohort B Group 2: Chlamydia trachomatis Seronegative (Experimental): Participants will receive three medium dose injections of Chlamydia mRNA Vaccine
  Interventions: Biological: Chlamydia mRNA Vaccine
- Sentinel Cohort C Group 3: Chlamydia trachomatis Seronegative (Experimental): Participants will receive three high dose injections of Chlamydia mRNA Vaccine
  Interventions: Biological: Chlamydia mRNA Vaccine
- Sentinel Cohort A, B and C Group 4: Chlamydia trachomatis Seronegative (Placebo Comparator): Participants will receive three injections of Placebo
  Interventions: Other: Placebo
- Sentinel Cohort A Group 5: Chlamydia trachomatis Seropositive (Experimental): Participants will receive three low dose injections of Chlamydia mRNA Vaccine
  Interventions: Biological: Chlamydia mRNA Vaccine
- Sentinel Cohort B Group 6: Chlamydia trachomatis Seropositive (Experimental): Participants will receive three medium dose injections of Chlamydia mRNA Vaccine
  Interventions: Biological: Chlamydia mRNA Vaccine
- Sentinel Cohort C Group 7: Chlamydia trachomatis Seropositive (Experimental): Participants will receive three medium dose injections of Chlamydia mRNA Vaccine
  Interventions: Biological: Chlamydia mRNA Vaccine
- Sentinel Cohort A, B and C Group 8: Chlamydia trachomatis Seropositive (Placebo Comparator): Participants will receive three injections of Placebo
  Interventions: Other: Placebo
- Main Cohort Group 9: Chlamydia trachomatis Seronegative (Experimental): Participants will receive three low dose injections of Chlamydia mRNA Vaccine
  Interventions: Biological: Chlamydia mRNA Vaccine
- Main Cohort Group 10: Chlamydia trachomatis Seronegative (Experimental): Participants will receive three medium dose injections of Chlamydia mRNA Vaccine
  Interventions: Biological: Chlamydia mRNA Vaccine
- Main Cohort Group 11: Chlamydia trachomatis Seronegative (Experimental): Participants will receive three high dose injections of Chlamydia mRNA Vaccine
  Interventions: Biological: Chlamydia mRNA Vaccine
- Main Cohort Group 12: Chlamydia trachomatis Seronegative (Placebo Comparator): Participants will receive three injections of Placebo
  Interventions: Other: Placebo
- Main Cohort Group 13: Chlamydia trachomatis Seropositive (Experimental): Participants will receive three low dose injections of Chlamydia mRNA Vaccine
  Interventions: Biological: Chlamydia mRNA Vaccine
- Main Cohort Group 14: Chlamydia trachomatis Seropositive (Experimental): Participants will receive three medium dose injections of Chlamydia mRNA Vaccine
  Interventions: Biological: Chlamydia mRNA Vaccine
- Main Cohort Group 15: Chlamydia trachomatis Seropositive (Experimental): Participants will receive three high dose injections of Chlamydia mRNA Vaccine
  Interventions: Biological: Chlamydia mRNA Vaccine
- Main Cohort Group 16: Chlamydia trachomatis Seropositive (Placebo Comparator): Participants will receive three injections of Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Chlamydia mRNA Vaccine — Pharmaceutical Form: Suspension for injection
  Route of Administration:
  Intramuscular injection
  Arms: Main Cohort Group 10: Chlamydia trachomatis Seronegative; Main Cohort Group 11: Chlamydia trachomatis Seronegative; Main Cohort Group 13: Chlamydia trachomatis Seropositive; Main Cohort Group 14: Chlamydia trachomatis Seropositive; Main Cohort Group 15: Chlamydia trachomatis Seropositive; Main Cohort Group 9: Chlamydia trachomatis Seronegative; Sentinel Cohort A Group 1: Chlamydia trachomatis Seronegative; Sentinel Cohort A Group 5: Chlamydia trachomatis Seropositive; Sentinel Cohort B Group 2: Chlamydia trachomatis Seronegative; Sentinel Cohort B Group 6: Chlamydia trachomatis Seropositive; Sentinel Cohort C Group 3: Chlamydia trachomatis Seronegative; Sentinel Cohort C Group 7: Chlamydia trachomatis Seropositive
Other: Placebo — Pharmaceutical Form:
  Solution for injection
  Route of Administration:
  Intramuscular injection
  Arms: Main Cohort Group 12: Chlamydia trachomatis Seronegative; Main Cohort Group 16: Chlamydia trachomatis Seropositive; Sentinel Cohort A, B and C Group 4: Chlamydia trachomatis Seronegative; Sentinel Cohort A, B and C Group 8: Chlamydia trachomatis Seropositive

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, and immunogenicity of different dose levels (low, medium, and high) of Chlamydia messenger ribonucleic acid (mRNA) Vaccine candidate in adult participants aged 18 to 29 years.

This study will consist of 3 Sentinel Cohorts and a Main Cohort, with the Sentinel Cohorts assessing the safety of the different dose levels in a stepwise manner.

All participants will be followed up to 12 months after the last study intervention administration. Thus, the expected duration of the participant's involvement will be 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 29 years on the day of inclusion
* New sex partner within the past 6 months, or more than one current sex partner, or partner with known previous or coexisting sexually transmitted infection (STI), or inconsistent condom use
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  * Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be surgically sterile.

OR

• Is of childbearing potential and agrees to use an effective contraceptive method from at least 4 weeks prior to study intervention administration until at least 4 weeks after the last study intervention administration.

* A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) at the screening visit and before each subsequent study intervention administration

Exclusion Criteria:

* Any screening laboratory parameter with laboratory abnormalities as per local reference range and that are greater than Grade 2 or deemed clinically significant in the opinion of the Investigator
* Participants who are Chlamydia trachomatis (CT) and/or Neisseria gonorrhea (NG) NAAT positive at screening visit
* Self-reported or documented seropositivity for HIV antigen and/or antibodies (Abs), hepatitis B virus surface antigen (HBsAg), hepatitis B core antibodies (HBcAbs), or hepatitis C virus (HCV) Abs infection at screening visit
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the study intervention components, or history of a life-threatening reaction to the study intervention(s) used in the study or to a product containing any of the same substances
* Previous history of myocarditis, pericarditis, and/or myopericarditis
* Known history of previous history of Guillain-Barre syndrome and other immune mediated demyelinating conditions that include but are not limited to Multiple Sclerosis (MS), Neuromyelitis Optica (NMO), acute disseminated encephalomyelitis (ADEM), Transverse myelitis
* Screening electrocardiogram (ECG) value that is consistent with possible myocarditis, pericarditis, and/or myopericarditis or screening ECG that demonstrates clinically relevant abnormalities, per investigator, that may affect participant safety or study results
* Self-reported thrombocytopenia, contraindicating intramuscular injection, based on investigator's judgment
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular injection, based on investigator's judgment
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Moderate or severe acute febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of study intervention administration. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion
* Receipt of any mRNA vaccine/product in the 2 months preceding study enrollment or planned receipt of any mRNA vaccine/product within the 2 months following any study intervention administration
* Receipt of any vaccine (other than the study vaccine) in the 4 weeks preceding any study intervention administration or planned receipt of any vaccine (other than the study vaccine) in the 4 weeks following any study intervention administration, except influenza which may be received at least 2 weeks before or 2 weeks after any study vaccination
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months

Note: The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1560 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2028-01-03 (Estimated); Study Completion 2028-01-03 (Estimated)

PRIMARY OUTCOMES:
Presence of immediate unsolicited systemic adverse events (AEs) | Within 30 minutes after each vaccine injection
  Number of participants with immediate unsolicited systemic adverse events (AEs) reported in the 30 minutes after each vaccine injection.
Presence of solicited injection site and systemic reactions | Up to 7 days after each vaccine injection
  Number of participants with solicited injection site and systemic reactions occurring up to 7 days after each vaccine injection.
Presence of unsolicited AEs | Up to 28 days after each vaccine injection.
  Participants with unsolicited AEs reported up to 28 days after each vaccine injection.
Presence of medically attended adverse events (MAAEs) | Up to 6 months after last vaccine injection
  Number of participants with MAAEs reported after each vaccine injection and up to 6 months after last vaccine injection.
Presence of all serious AEs (SAEs) and all adverse events of special interest (AESIs) | Up to 12 months after last vaccine injections
  Number of participants with SAEs and all AESIs reported after each vaccine injection and up to 12 months after last vaccine injection
Presence of related SAEs, and fatal SAEs | Throughout the study, appriximatley 18 months
  Number of participants with related SAEs, and fatal SAEs throughout the study
Presence of out-of-range biological test results (Sentinel Cohort and Safety Subset of Main Cohort) | Up to 7 days after each vaccination injections
  Number of participants with out-of-range biological test results up to 7 days after each vaccine injection

SECONDARY OUTCOMES:
Assessment of serum binding antibodies to specific Chlamydia trachomatis antigens and whole bacteria in immunogenicity subset | Before each vaccine injection through 1 month after each vaccine injection
  Binding Immunoglobulin (Ig) will be measured using a multiplex electrochemiluminescent (ECL) based binding assay
Geometric mean cell-mediated immune response of antigen-specific T helper type 1 (Th1) and T helper type 2 (Th2) cytokine-producing T cells by phenotype | Before each vaccine injection through 1 month after each vaccine injection
  Geometric mean cell-mediated immune responses will be measured by an intracellular cytokine staining assay over time

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (6):
  - Investigational Site Number : 0360002, Bruce, Australian Capital Territory
  - Investigational Site Number : 0360006, Maroubra, New South Wales
  - Investigational Site Number : 0360005, Sydney, New South Wales
  - Investigational Site Number : 0360001, Albion, Queensland
  - Investigational Site Number : 0360004, Morayfield, Queensland
  - Investigational Site Number : 0360003, Southport, Queensland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org